CLINICAL TRIAL: NCT05178862
Title: A Phase 3, Multicenter, Prospective, Randomized, Double-blind Study of Two Treatment Regimens for Candidemia and/or Invasive Candidiasis: Intravenous Echinocandin Followed by Oral Ibrexafungerp Versus Intravenous Echinocandin Followed by Oral Fluconazole (MARIO)
Brief Title: A Phase 3, Randomized, Double-blind Study for Patients With Invasive Candidiasis Treated With IV Echinocandin Followed by Either Oral Ibrexafungerp or Oral Fluconazole
Acronym: MARIO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination is not related to safety or efficacy concerns for Ibrexafungerp. GSK's decision is to focus efforts and resources on commercialization of Ibrexafungerp for the already approved VVC and rVVC indications.
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCY-078-302; MSG-20 (Other: Mycoses Study Group (MSGERC))
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Candidiasis, Invasive; Candidemia
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia | interventions — ibrexafungerp; Fluconazole; Echinocandins; Caspofungin; Micafungin; Anidulafungin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV echinocandin followed by oral ibrexafungerp (SCY-078) (Experimental)
  Interventions: Drug: SCY-078; Drug: Echinocandin
- IV echinocandin followed by oral fluconazole (Active Comparator)
  Interventions: Drug: Fluconazole; Drug: Echinocandin

INTERVENTIONS:
Drug: SCY-078 — Oral ibrexafungerp (SCY-078) as step-down therapy.
  Other Names: Ibrexafungerp
  Arms: IV echinocandin followed by oral ibrexafungerp (SCY-078)
Drug: Fluconazole — Oral fluconazole (SCY-078) as step-down therapy.
  Other Names: Diflucan
  Arms: IV echinocandin followed by oral fluconazole
Drug: Echinocandin — Intravenous echinocandin
  Other Names: Caspofungin; Micafungin; Anidulafungin

SUMMARY:
This is a multicenter, randomized, double-blind study of two treatment regimens for invasive candidiasis included candidemia. Subjects will receive intravenous echinocandin followed by oral ibrexafungerp (SCY-078) vs intravenous echinocandin followed by oral fluconazole.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject is a male or female adult ≥ 18 years of age on the day the study informed consent is signed.
* Subject has a diagnosis of candidemia and/or invasive candidiasis, defined as evidence of Candida spp in either a bloodstream or tissue culture from a normally sterile site (excluding eye, cardiac tissue, bone tissue, central nervous system or prosthetic device) collected ≤ 4 days (within 96 hours) prior to initiation of IV echinocandin accompanied by any related clinical signs and/or symptoms (e.g., fever [on one occasion > 38°C], hypotension, or local signs of inflammation).

Key Exclusion Criteria:

* Subject has any of the following forms of invasive candidiasis at Screening:

  * Septic arthritis in a prosthetic joint (septic arthritis in a native joint is allowed),
  * Osteomyelitis,
  * Endocarditis or myocarditis,
  * Meningitis, endophthalmitis, or any central nervous system infection,
  * Chronic disseminated candidiasis,
  * Urinary tract candidiasis due to ascending Candida infection secondary to unresolved obstruction or non-removeable device in the urinary tract,
  * Patients with a sole diagnosis of mucocutaneous candidiasis, i.e., oropharyngeal, esophageal, or genital candidiasis; or Candida lower urinary tract infection or Candida isolated solely from respiratory tract specimens,
  * Patients with concurrent invasive fungal infection other than Candida spp., e.g., cryptococcosis, mold infection or endemic fungal infection,
  * Patients who failed a previous antifungal therapy for the same infection,
  * Subject has an inappropriately controlled fungal disease source (e.g., indwelling vascular catheter or device that cannot be removed or an abscess that cannot be drained) that is likely to be the source of the candidemia or invasive candidiasis.
* Subject has abnormal liver test parameters: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels > 10-fold the upper limit of normal (ULN).
* Subject has severe hepatic impairment and a history of chronic cirrhosis (Child-Pugh score > 9).
* Subject has received more than 48 hours of non-echinocandin antifungal therapy for the treatment of invasive candidiasis (including candidemia) within 96 hours preceding initiation of IV echinocandin.

  o Exception: Receipt of antifungal therapy to which any Candida spp. isolated in qualifying culture is not susceptible.
* Baseline QTcF ≥ 500 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
All-cause mortality (US FDA Only) | Day 30
  The number and percentage of subjects in each treatment group who are alive and deceased in the ITT population.
Global Response at End of Treatment (EU European Medicines Agency [EMA] Only) | Up to 6 weeks
  The percentage of subjects with Successful Global Response, as determined by the Data Review Committee

SECONDARY OUTCOMES:
Global Response at Day 14 | Day 14
  The percentage of subjects with Successful Global Response, as determined by the Data Review Committee

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (101):
- United States (26):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Banner University Medical Center-Tucson, Tucson, Arizona
  - UC Davis Medical Center, Sacramento, California
  - UCSF School of Medicine, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Denver, Colorado
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - LSU Health Sciences Center, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Duke University, Durham, North Carolina
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (3):
  - Saint Luc University Hospital, Brussels
  - University Hospital Ghent, Ghent
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
- Bulgaria (3):
  - University Multiprofile Hospital for Active Treatment "Eurohospital Plovdiv", Plovdiv, Department of Surgery, Plovdiv
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Clinic of Purulent-Septic Surgery, Sofia
  - University Multiprofile Hospital for Active Treatment "Prof. Dr. Stoyan Kirkovich", Stara Zagora
- Canada (3):
  - Princess Margaret Hospital, Toronto, Ontario
  - University Health Network- Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- China (21):
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guandong, Guangzhou
  - The First Affiliated Hospital of Jinan University, Guandong, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangdong, Guangzhou
  - The Third Affiliated Hospital Of Sun Yat-Sen University (ZSSY), Guangdong, Guangzhou
  - Hainan General Hospital, Haikou, Hainan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Liuzhou People's Hospital, Liuchow, Liuzhou
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Institute of Antibiotics, Shanghai, Shanghai Municipality
  - Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Chinese Academy of Medical Sciences, Jinghai, Tianjin Municipality
  - Tianjin Medical University General Hospital, Xiaobailou, Tianjin Municipality
  - The First Hospital of Kunming, Kunming, Yunnan
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Yuzhong
  - The first affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincal Hospital of Chinese Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Affiliated to Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Lishui People's Hospital, Lishui, Zhejiang
- France (5):
  - Victor Dupouy Hospital Center Argenteuil, Argenteuil
  - Nantes University Hospital Center, Nantes
  - Paris University Hospitals Center- Cochin Hospital, Paris
  - Saint-Louis Hospital, Paris
  - University Hospital Center of Poitiers, Poitiers
- Germany (6):
  - University Hospital Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Univeristy Hospital Jena, Jena, Thuringia
  - University Hospital Cologne, Cologne
  - Frankfurt University Clinic, Frankfurt
  - Municipal Hospital Munich GMbH/Hospital Neuperlach, Munich
  - Helios Clinic Wuppertal, Wuppertal
- Greece (5):
  - General Hospital of Athens "Evangelismos", 1st Department of Critical Care, Athens
  - General Hospital of Athens "Evangelismos", Athens
  - LAIKO General Hospital, Athens
  - University General Hospital "Attikon", Athens
  - General Hospital of Thessaloniki "Ippokratio", Thessaloniki
- Israel (4):
  - Lady Davis Carmel Medical Center, Infectious Diseases Unit, Haifa
  - Rambam Health Care Campus, Institute of Infectious Diseases, Haifa
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (4):
  - IRCCS- University Hospital San Martino-IST, Genoa, Liguria
  - Big Metropolitan Hospital Niguarda Regional Health Authority, Milan
  - University Polyclinic Hospital of Modena, Modena
  - Central Friuli University Healthcare Company, Udine
- South Africa (7):
  - Lakeview Hospital, Benoni, Gauteng
  - Netcare Jakaranda Hospital, Pretoria, Gauteng
  - Zuid-Afrikaans Hospital, Pretoria, Gauteng
  - Life Groenkloof Hospital, Pretoria, Gauteng
  - FCRN Clinical Trials Centre, Vereeniging, Gauteng
  - Mediclinic Victoria, Tongaat, KwaZulu-Natal
  - University of Pretoria and Steve Biko Academic Hospital, Pretoria
- South Korea (5):
  - Keimyung University - Dongsan Medical Center, Daegu
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Gangnam Severance Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Spain (9):
  - University Hospital Virgen Macarena, Seville, Andalusia
  - Hospital Clínic de Barcelona, Barcelona, Catalonia
  - Hospital del Mar Medical Research Institute (IMIM), Barcelona, Catalonia
  - University Hospital Ramon y Cajal, Madrid
  - General University Hospital Gregorio Maranon, Madrid
  - University Hospital de La Princesa, Madrid
  - University Hospital Puerta de Hierro Majadahonda, Madrid
  - University and Polytechnic Hospital La Fe, Valencia
  - University Clinical Hospital of Valencia, Valencia